CLINICAL TRIAL: NCT00915447
Title: Diesel Exhaust Particles and Leukotriene Production
Status: Withdrawn | Type: Observational
Why Stopped: Investigator left the institution prior to enrollment of first participant
Sponsor: University of California, Los Angeles (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB # 07-10-025; FAU # 441329-ZC-77586
Record Dates: First submitted 2009-06-05; First posted 2009-06-08 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Allergic Rhinitis
Keywords: Cat Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine, Nasal Lavage

GROUPS / COHORTS (1):
- Cat Allergic Rhinitis: Individuals with cat allergic rhinitis, yet without routine cat exposure

SUMMARY:
The purpose of this study is to measure the effects of allergens and/or diesel exhaust particles in the nose to learn more about allergic responses in individuals with cat allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 65 years old.
2. Positive prick (epicutaneous) skin test to standardized cat with a wheal equal to or greater than 3 mm and with a surrounding flare.
3. Ability to give informed consent.

Exclusion Criteria:

1. Pregnancy or breast-feeding. (Pregnancy and the period during breast feeding can affect nasal congestion and be a confounder in this regard.)
2. Systemic corticosteroid use within the previous three months or anytime during the challenge protocol.
3. Topical nasal corticosteroid use within the past month or anytime during the challenge protocol.
4. Systemic antihistamines or decongestant use within past two weeks or anytime during the trial.
5. Chronic sinusitis or chronic non-allergic rhinitis.
6. Use of reserpine.
7. Cigarette smoking within the past year or during the challenge protocol
8. Use of topical nasal antihistamines, chromoglycolates (chromolyn, Cromlon®), decongestants or non-steroidal anti-inflammatory agents (NSIADS) within the preceding week or anytime during the challenge protocol.
9. Present or treatment within the past 10 years with allergy immunotherapy (injections).
10. Present or past treatment with anti-IgE therapy.
11. Any unusual exposure to air pollutants (e.g., working as a diesel mechanic) that, in the opinion of the investigators, might compromise the individual's ability to participate in the study.
12. Living arrangement where the subject has a cat dwelling within the subject's habitation.
13. Any serious heart, lung, neurological or kidney disease that in the opinion of the investigators would impair the individual's ability to participate in the study.
14. Use of asthma-required medications.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-04 (Actual); Primary Completion 2013-04-11 (Actual); Study Completion 2013-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Riedl, M.D., M.S., Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States